CLINICAL TRIAL: NCT01197742
Title: Sweetheart: Risiko-Management Von Diabetikern Mit Akutem Myokardinfarkt
Brief Title: Sweetheart-Register: Risk Management of Diabetics with Acute Myocardial Infarction
Acronym: Sweetheart
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: Sweetheart
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Diabetes; STEMI; NSTEMI; Myocardial Infarction
Keywords: Diabetes; STEMI; NSTEMI; Myocardial infarction
MeSH Terms: conditions — Diabetes Mellitus; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Sweetheart register (Risk management of Diabetics with acute myocardial infarction) documents both the prevalence of pathologic glucose metabolism in consecutive high-risk patients with STEMI and NSTEMI in daily hospital routine as well as the anti-diabetic acute and long-term therapy. Furthermore the register will provide data about the implementation of new guidelines for the interventional and adjuvant medical therapy of STEMI and NSTEMI.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients with acute (no older than 24 h) ST-Elevation Myocardial infarction
* consecutive patients with acute (no older than 24 h) Non-ST-Elevation Myocardial infarction

Exclusion Criteria:

* missing informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all consecutive patients with acute (no older than 24 h) ST-Elevation Myocardial infarction or acute (no older than 24 h) Non-ST-Elevation Myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 2772 (Actual)
Dates: Start 2007-04-20 (Actual); Primary Completion 2009-10-05 (Actual); Study Completion 2009-10-05 (Actual)

PRIMARY OUTCOMES:
Documentation of the characteristics consecutive patients with acute STEMI or NSTEMI in daily hospital routine in Germany | 04/01/2007-09/30/2009

SECONDARY OUTCOMES:
Documentation of the fraction of patients with (I) a previous know Diabetes Mellitus (DM) type I and II, (II) a newly diagnosed DM, (III) diagnosed with IFG or IGT for the first time | 04/01/2007-09/30/2009
Documentation of acute invasive and adjuvant medicamentous therapy of STEMI and NSREMI in hospital daily routine in Germany | 04/01/2007-09/30/2009
Documentation of diabetic therapy during the acute phase of a myocardial infarction | 04/01/2007-09/30/2009
Documentation of the hospital mortality, the serious but non-fatal complications (stroke, re-myocardial infarction) and other bleeding complications | 04/01/2007-09/30/2009
Verification of the implementation of a therapy according to the guidelines for STEMI / NSTEMI in daily hospital routine | 04/01/2007-09/30/2009

CONTACTS AND LOCATIONS:
Overall Officials: Anselm K Gitt, MD, Study Chair — Stiftung Institut für Herzinfarktforschung; Jochen Senges, MD, Study Chair — Stiftung Institut für Herzinfarktforschung
Locations (2):
- Germany (2):
  - Städ Krankenhaus münchen Schwabing, München
  - Klinikum Nürnberg Süd /Cardiology, Nuremberg